CLINICAL TRIAL: NCT02964650
Title: The Safety and Efficacy of Optimising Pacemaker Heart Rate for Contractility: Effects on Walk Time, Cardiac Remodelling and Quality of Life.
Brief Title: Optimising Pacemaker Therapy for Contractility
Acronym: OPT-C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, KK Witte, Senior Lecturer in Cardiology, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRAS 218963
Record Dates: First submitted 2016-11-08; First posted 2016-11-16 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard rate-response settings (No Intervention): Patients allocated to standard rate-response settings.
- Personalised rate-response settings (Experimental): Patients allocated to optimised rate-response settings.
  Interventions: Device: Personalised rate-response settings

INTERVENTIONS:
Device: Personalised rate-response settings — Rate response range fixed to limits suggested by force-frequency curve
  Arms: Personalised rate-response settings

SUMMARY:
The investigators have demonstrated that they can reliably identify an optimum heart rate range for contractility of the left ventricle in patients with chronic heart failure (CHF). They have also demonstrated in an acute cross-over study that keeping the heart rate in this range (versus standard rate-response programming) in patients with CHF is associated with increased exercise time on a treadmill (around 60s or 10%). They now want to explore in a randomised, placebo-controlled trial whether optimal programming versus standard rate-response programming for 6 months leads to appreciable improvements in exercise time and quality of life, while having no adverse effects on left ventricular function and battery longevity.

60 patients with CHF and a pacemaker will undergo the non-invasive echocardiographic assessment to establish the force frequency relationship and the optimal heart rate for contractility. They will then perform a treadmill walk test and fill out a quality of life questionnaire. They will then be randomised to optimal rate-response settings or standard rate response settings and followed up at 6 months at which point the tests will be repeated.

DETAILED DESCRIPTION:
Design: This will be a randomised, double-blind 'placebo' controlled trial of optimised programming versus standard rate-response settings, aiming to determine whether the short term improvements translate into longer term benefits.

Study participants: 60 adult patients (>18years) aiming for 50 matched datasets (25 in each arm).

Study Procedures: Patients attending the heart failure clinic, the pacemaker clinic or previous participants in the acute cross-over study (pilot data 2) will be approached with a standard letter and information sheet and then a telephone call to make sure any remaining questions are answered.

Patients agreeing to participate will attend the clinical research facility (CRF) and will be asked to sign a consent form. Each patient will have a standard device check, check of their demographic data, and co-morbidities. The investigators will record a resting cardiac ultrasound, and, in those who did not participate in the pilot study (or did so more than six months previously), we will measure the force frequency relationship (FFR) as described to determine critical heart rate (HR), and the optimal range of HR rise. All images will be stored for offline analysis. Participants will then be asked to do a symptom-limited walk test on the treadmill (until they cannot do any more). At this first visit, participants will also complete a quality of life questionnaire. All of these activities will take place in the Clinical Research Facility at Leeds General Infirmary.

Randomisation: Each patient will then be randomised to either optimised programming (n=30) as predicted by their force-frequency curve or standard settings (n=30). In the optimised group, programming will keep heart rates below the critical HR. Randomisation will be by a random number generator and programming will be undertaken by one of my colleagues to maintain blinding.

Follow-up: Each patient will be called at one month to check that they are tolerating any changes and will then be invited back at 6 months for a repeat resting echocardiogram, treadmill walk test and quality of life assessment.

Data: All data will be stored on a bespoke Excel spreadsheet on an LTHT server in a password-protected folder.

Primary Endpoint: The effects of heart rate programming that optimises heart rate for contractility on change in treadmill-based walk distance over six months in patients with heart failure and a pacemaker.

Secondary endpoints: 1) the safety of pacemaker programming optimised for heart rate in patients with heart failure and a pacemaker, 2) the effect of this programming on change of quality of life at 6 months 3) the effect of this programming on change in cardiac function at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic CHF due to left ventricular systolic dysfunction (LVEF<45%),
* Cardiac pacemaker,
* Able to perform a peak exercise test,
* Willing and able to give informed consent.

Exclusion Criteria:

* Angina pectoris symptoms limiting exercise tolerance,
* Unstable heart failure symptoms (medical therapy changes in last three months), Poor image quality,
* Calcium channel blockers (CCBs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Treadmill walk time | 6 months
  Time walked during a standard incremental treadmill test

SECONDARY OUTCOMES:
Quality of life | 6 months
  EQ5D-5L
Left ventricular function by echocardiography | 6 months
Battery longevity | 6 months
  Measured in years remaining at current settings

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Witte, MD, Principal Investigator — University of Leeds
Locations (1):
- Leeds General Infirmary, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gierula J, Lowry JE, Paton MF, Cole CA, Byrom R, Koshy AO, Chumun H, Kearney LC, Straw S, Bowen TS, Cubbon RM, Keenan AM, Stocken DD, Kearney MT, Witte KK. Personalized Rate-Response Programming Improves Exercise Tolerance After 6 Months in People With Cardiac Implantable Electronic Devices and Heart Failure: A Phase II Study. Circulation. 2020 May 26;141(21):1693-1703. doi: 10.1161/CIRCULATIONAHA.119.045066. Epub 2020 Apr 17. PMID 32299222